CLINICAL TRIAL: NCT06555666
Title: Practice of Scuba Diving by as Many People as Possible: Effect of Medical Assessment to Provide a Suitable and Individualised Framework for Practice
Brief Title: Practice of Scuba Diving by as Many People as Possible: Effect of Medical Assessment to Provide a Suitable and Individualised Framework for Practice (Plongée Santé)
Acronym: Healthy-diving
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0226 - Healthy diving
Record Dates: First submitted 2021-11-08; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2023-08

CONDITIONS: Diving Barotrauma
Keywords: scuba diving; medical fitness; sport for health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study focuses on the practice of recreational scuba diving by people who have obtained medical advice for their practice in the hyperbaric and underwater medicine department of the Brest University Hospital. These people may have no health problem or on the contrary consult because they have a pathology and want a medical advice on the impact of this health problem on their practice: this is the case for about the half of these consultants.

For the latter, there are no data concerning the relevance of a medical advice response and a proposal for an appropriate technical practice framework (restriction of dive depth, duration, etc.). A relevant answer results in a practice without diving accidents or decompensation of the pathology and a decision accepted and respected by the practitioner.

This study aims to analyze the state of health of the service's consultants and medical recommendations formulated at the end of this consultation, by retrospective analysis of the consultation files, and to interview the consultants on their practice of diving, their state of health and any problems encountered since their consultation.

The purpose is to validate the hypothesis that a practice of underwater diving is possible and beneficial, with an acceptable risk in case of a risk factor or pathology using a framework of advice and restrictions of adapted and individualized practice ("sport for health").

DETAILED DESCRIPTION:
This is a single-center retrospective study on health data. The methodology includes a collection of data on health and practice of scuba diving, figuring on the medical consultation files and then carrying out a telephone interview of people seen in diving medicine consultation between 01/01/2015 and on 12/31/2018 in the hyperbaric and underwater medicine department of the Brest University hospital.

One month before the start of these interviews, an information letter on the study is sent by post, giving the possibility of opposing it.

The main evaluation criteria are the number of dives carried out since the consultation (and the average number of dives per year of practice), and the number of accidents or incidents during the practice of recreational scuba diving in the framework proposed, during the months or years following the medical consultation The secondary evaluation criteria are the evolution of the chronic pathology, the evolution of health status in general, the number of hours of practice of a physical and sport activity per week, the respect of the technical practice framework recommended.

ELIGIBILITY:
Inclusion Criteria:

* People who asked for a medical advice for the diving practice in a consultation in the hyperbaric and underwater medicine department of the Brest University hospital from 2015/01/01 to 2018/12/31

Exclusion Criteria:

* refusal

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The population include new potential divers and confirmed divers who asked for a medical advice about their practice of diving.
  About a half of this population have had a diving injury or has a chronic pathology.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
injury during diving practice since the consultation | 1 month
  type and number of diving injury

SECONDARY OUTCOMES:
evolution of health status | 1 month
  qualitative scale : new pathology, worse, stable or better
evolution of the chronic pathology | 1 month
  qualitative scale : worse, stable, recurrence or remission
duration of physical or sport practice per week | 1 month
  in hours per week
medical recommendation respect | 1 month
  for each participant, comparison between the medical recommended practice framework and the actual practice declared; then percentage of participant that indicate following the medical recommendation
number of dives carried out since the consultation | 1 month
  average number per year of practice

CONTACTS AND LOCATIONS:
Overall Officials: Anne HENCKES, Principal Investigator — CHRU Brest
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three months and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.